CLINICAL TRIAL: NCT04213300
Title: The Association Between a Low Carbohydrate Diet, Glycaemic Control and Quality of Life in Australian Adults Living With Type 1 Diabetes Mellitus: A Pilot Study
Brief Title: Low Carbohydrate Diet, Glycaemic Control and Quality of Life in Australian Adults With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Gold Coast Hospital and Health Service (Other Government)
Collaborators: University of Canberra (Other)
Responsible Party: Sponsor
Other Study IDs: HREC/2019/QGC/54049
Record Dates: First submitted 2019-11-27; First posted 2019-12-30 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Quality of life; Glycaemic control; Low carbohydrate diet
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low carbohydrate dietary group: Participants n = 23
  Participants:
  * Male, female or unspecified gender;
  * 18 years of age or over;
  * Type 1 diabetes for ≥1 year from diagnosis date and
  * Individuals who administer insulin using multiple daily injections.
  Interventions: Other: Low carbohydrate diet

INTERVENTIONS:
Other: Low carbohydrate diet — Study duration: 13 weeks (run in phase = 1 week; low carbohydrate diet phase = 12 weeks).
  Each participant will be provided with an individualised meal plans to meet their energy needs as per the Schofield formula and a macronutrient distribution of 20% for carbohydrate, 25% for protein and 55% for fat.
  Participants will self-report quality of life using a validated diabetes specific quality of life questionnaire for Australian adults and HbA1c (pre and post intervention phase of 13 weeks duration) .

SUMMARY:
The aim of this study is to examine the association between a low carbohydrate diet, quality of life and glycaemic control in Australian adults with T1DM. The first phase of the study will develop and validate a diabetes specific quality of life questionnaire for adults with T1DM. The second phase will undertake a low carbohydrate diet intervention and examine its association with quality of life and glycaemic control, pre and post the dietary intervention. The novel outcomes will include a new validated Australian T1DM specific quality of life questionnaire and an investigation as to whether a low carbohydrate diet mediates the relationship between quality of life and glycaemic control in Australian adults with T1DM.

DETAILED DESCRIPTION:
Phase 1:

Aim: To develop a reliable and valid diabetes specific quality of life questionnaire for use in Australian adults living with type 1 diabetes mellitus (T1DM).

Objectives:

1. To develop a new Australian diabetes specific quality of life online questionnaire integrating participant feedback using a one to one interview method;
2. Pilot the study developed online questionnaire with adults that have type 1 diabetes mellitus and
3. Conduct factorial validation of the study developed online questionnaire using advanced statistical modelling techniques.

Phase 2:

Aim: The aim of this study is to examine the association between a low carbohydrate diet, quality of life and glycaemic control in adults living with T1DM.

Objectives:

1. To examine the association between quality of life and glycaemic control in adults with T1DM;
2. Implement a low carbohydrate diet in a cohort of adults living with T1DM;
3. Examine the association between a low carbohydrate diet and glycaemic control in adults with T1DM: pre and post intervention;
4. Examine the association between quality of life and a low carbohydrate in adults with T1DM: pre and post intervention and
5. Investigate whether a low carbohydrate diet mediates the relationship between quality of life and glycaemic control in adults with T1DM.

ELIGIBILITY:
Inclusion Criteria:

* Male, female or unspecified gender;
* 18 years of age or over;
* Type 1 diabetes for ≥1 year from diagnosis date and
* Individuals who administer insulin using multiple daily injections.

Exclusion Criteria:

* Patients with type 2 diabetes mellitus;
* Patients with gestational diabetes mellitus;
* Presence of a known food allergy or intolerance that may affect the participants' health or adherence during the intervention;
* History of an eating disorder;
* BMI <25.0kg/m2 to 29.9kg/m2;
* Age <18 years;
* An active medical problem that may hinder the persons' ability to take part or potentially affect study outcomes e.g. a recent myocardial infarction, stroke or peripheral revascularisation (within 3 months), active treatment of diabetic retinopathy, recent serious infection (requiring in-hospital treatment or prolonged antibiotic therapy), active mental health complaint or other active medical problems determined by medical staff;
* Pregnancy or expectation of conceiving. Participants will be withdrawn at any stage from the study if pregnancy occurs;
* The use of medications that may affect body weight/body composition (including but not limited to phentermine and corticosteroids);
* Those for whom the written materials may be unsuitable such as vision impaired or illiterate individuals;
* Those unable to understand English;
* Those who failed to provide informed consent and
* Those who administer insulin using a continuous subcutaneous insulin infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Male, female or unspecified gender;
  * 18 years of age or over;
  * Type 1 diabetes for ≥1 year from diagnosis date and
  * Individuals who administer insulin using multiple daily injections.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Self reported quality of life at baseline pre intervention | Baseline (pre intervention)
  Baseline (pre intervention) participant self reported quality of life using the newly validated Australian diabetes specific quality of life questionnaire which uses a Likert scale of 1 = very strongly disagree to 10 = very strongly agree, from baseline to 12 weeks after intervention
Self reported quality of life at 12 weeks post intervention | 12 weeks (post intervention)
  % change in participant self reported quality of life from baseline to 12 weeks (post intervention) using the newly validated Australian diabetes specific quality of life questionnaire which uses a Likert scale of 1 = very strongly disagree to 10 = very strongly agree, from baseline to 12 weeks after intervention
Glycaemic control (HbA1c) at baseline pre intervention | Baseline (pre intervention)
  Baseline (pre intervention) in glycaemic control (HbA1c)
Glycaemic control (HbA1c) | 12 weeks (pre and post intervention)
  % change in glycaemic control from baseline to 12 weeks (post intervention) (HbA1c)

CONTACTS AND LOCATIONS:
Overall Officials: Janine Paul, MSc, Principal Investigator — Gold Coast Hospital and Health Service
Locations (1):
- Gold Coast Hospital and Health Service, Gold Coast, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
The data collected in this study is specific to this doctoral research project. Therefore, there will be no data sharing with any other researchers who are not members of this study. Where a current research team member wishes to use any of this data research purposes, the research must be approved by an Ethics committee, involve the PI who will ultimately retain oversight of all future uses of data and will remain the ongoing custody of data and/or research outputs.

REFERENCES:
- [Derived] Paul J, Jani R, Davoren P, Knight-Agarwal C. Association Between a Low Carbohydrate Diet, Quality of Life, and Glycemic Control in Australian Adults Living With Type 1 Diabetes: Protocol for a Mixed Methods Pilot Study. JMIR Res Protoc. 2021 Mar 26;10(3):e25085. doi: 10.2196/25085. PMID 33769300